CLINICAL TRIAL: NCT01589159
Title: A Phase Ⅱ Study of an All-Oral Combination of Low-dose Etoposide/Capecitabine in Patients With Metastatic Breast Cancer Previously Treated With Anthracyclines and/or Taxanes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tao OUYANG (Other)
Responsible Party: Sponsor-Investigator, Tao OUYANG, Chairman of Breast Center, Peking University
Organization: Peking University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCP09
Record Dates: First submitted 2012-04-28; First posted 2012-05-01 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental)
  Interventions: Drug: Capecitabine; Drug: Etoposide

INTERVENTIONS:
Drug: Capecitabine — Drug:capecitabine 700mg/m2, twice daily on days 1-14.
Drug: Etoposide — Etoposide 30mg/m2, once daily on days 1-7.

SUMMARY:
This is a single-center, open-lable, non-comparative, prospective, phase Ⅱ efficacy and safety study. Eligible patients are enrolled in a single group. The investigators propose to determine the efficacy and safety of low-dose metronomic chemotherapy with Etoposide/Capecitabine in Patients with Metastatic Breast Cancer Previously Treated with Anthracyclines and/or Taxanes.

ELIGIBILITY:
Inclusion Criteria:

* female patients between 18 and 65 years old
* patients with metastatic breast cancer previousely treated with A/T
* able and willing to give consent to participate in the study

Exclusion Criteria:

* pregnant or lactating females
* other tumor history
* instable complication (e.g., myocardial infarction within 6 months,arrhythmia, unstable diabetes, hypercalcemia) or uncontrolled infection
* concurrent disease or condition that would make the patient inappropriate for study participation
* resist to participate in the study

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Clinical benefit rate | 24 weeks after the treatment
  Clinical benefit is defined as CR, PR, SD≥24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wei, Doctor, Study Chair — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality, China